CLINICAL TRIAL: NCT01309308
Title: The Impact of Sweeping the Membranes on Cervical Length and Labor: A Randomized Clinical Trial
Brief Title: Sweeping the Membranes, Cervical Length and Duration of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huriye Ayse Parlakgumus (Other)
Collaborators: Baskent University (Other)
Responsible Party: Sponsor-Investigator, Huriye Ayse Parlakgumus, MD, Baskent University
Organization: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KA 09/248
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Results first posted 2011-10-03 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Disorder of Amniotic Cavity and/or Membrane
Keywords: cervical length; sweeping the membranes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- The membranes swept group (Experimental): This group will have a sweeping of the membranes after the 38th of gestation at hospital, in order to reduce the latency period until labor. Sweeping of the membranes is done by the insertion of examiners finger between the decidua and fetal membranes and by the circular movement of the finger, the membranes are detached from the decidua.
  Interventions: Procedure: sweeping the membranes
- No sweeping group (Sham Comparator): This group will not have sweeping of the membranes, will only have vaginal ultrasound
  Interventions: Other: No sweeping group

INTERVENTIONS:
Procedure: sweeping the membranes — The cervical length will be measured and the patient will be examined to determine the Bishop score. Later the the membranes will be swept.
  Other Names: stripping the membranes; digital examination
  Arms: The membranes swept group
Other: No sweeping group — Cervical length will be measured by transvaginal USG and the patient will be examined to determine the Bishop score.
  Other Names: bishop score; digital examination
  Arms: No sweeping group

SUMMARY:
Sweeping the membranes in term pregnancy may shorten the cervix and reduce the time to delivery.

DETAILED DESCRIPTION:
Cervical length will be measured in both groups. The membranes will be swept in pregnancies beyond 38 weeks by digital examination in the study group. The control group will only be examined for Bishop score. Two days later cervical length will be Measured once more.

ELIGIBILITY:
Inclusion Criteria:

* The patients who completed the 38th week of pregnancy, otherwise healthy gravida who have no contraindication to vaginal delivery.

Exclusion Criteria:

* Women who have chronic disease complicating pregnancy, multiple pregnancies and in whom vaginal delivery is contraindicated.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huriye A Parlakgumus, MD, Principal Investigator — Baskent University
Locations (1):
- Baskent Universitesi Seyhan Arastirma ve Uygulama Hastanesi, Adana, Turkey (Türkiye)

REFERENCES:
- [Derived] Parlakgumus HA, Yalcinkaya C, Haydardedeoglu B, Tarim E. The impact of sweeping the membranes on cervical length and labor: a randomized clinical trial. Ginekol Pol. 2014 Sep;85(9):682-7. PMID 25322540

RESULTS

PARTICIPANT FLOW:
Recruitment Details: february-March 2011- department of obstetrics and gynecology
Pre-assignment Details: The participants are excluded from the study after assignment to the groups if they did not attend the second ultrasound measurement or if they delivered in another clinic.
Groups:
- The Membranes Swept Group: The patient whose amniotic membranes are detached by the circular movements of the examining fingers
- No Sweeping Group: The patients who did not have sweeping of the membranes
Period: Overall Study
Arm/Group | The Membranes Swept Group | No Sweeping Group
Started | 75 | 75
Completed | 69 | 71
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The Membranes Swept Group | No Sweeping Group | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 75 | 150
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.25 (5.06) | 28.11 (4.78) | 27.69 (4.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 75 | 150
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Cervical Shortening
Description: Cervix 1 was measured at the sagittal plane of cervix from external to the internal os. Two days later cervix 2 was measured the same way. The cervical shortening was calculated from subtracting cervix 1 from cervix 2.
Time Frame: 2days
Population: analysis was per person who delivered
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Sweeping: In women who had completed 38 weeks of gestation sweeping was performed by separating the lower membranes as much as possible from their cervical attachment, with three circumferential passes of the examining fingers for only once.
- Not Swept: Patients whose membranes are not swept
Arm/Group | Sweeping | Not Swept
Number analyzed (Participants) | 69 | 71
millimeters
  cervix1 | 27.45 (8.39) | 29.61 (8.97)
  cervix2 | 23.30 (8.84) | 23.88 (8.52)
  cervical shortening | 5.15 (4.42) | 5.72 (4.37)

2. Secondary Outcome: The Duration of Latency Until Labor
Description: The period (in days) from the last cervical measurement to the start of second phase of labor.
Time Frame: 15 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sweeping | Not Swept
Number analyzed (Participants) | 69 | 71
days | 6.33 (4.57) | 5.69 (4.11)

ADVERSE EVENTS:
Arm/Group | The Membranes Swept Group | No Sweeping Group
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

LIMITATIONS AND CAVEATS:
Patients who did not attend the second examination, patients who did not deliver in our clinic are excluded

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes